CLINICAL TRIAL: NCT02228395
Title: A Phase 1, Randomized, Subject- And Investigator-blind, Sponsor Open, Placebo Controlled, Single Ascending Dose Escalation Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Pf-04958242 Following Oral Dose Capsules in Healthy Subjects
Brief Title: Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Single Doses Of PF-04958242 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1701016; SAD-MAD (Other: Alias Study Number)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Single ascending doses; pharmacokinetics; safety; tolerability; healthy volunteers; cognitive impairment associated with schizophrenia (CIAS)
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Participants received 1 single dose of placebo, PF-04958242 0.6 mg, and PF-04958242 0.8 mg orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
  Interventions: Drug: PF-04958242; Drug: Placebo
- Cohort 2 (Experimental): Participants received 1 single dose of PF-04958242 0.35 mg, placebo, and PF-04958242 0.8 mg orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
  Interventions: Drug: PF-04958242; Drug: Placebo
- Cohort 3 (Experimental): Participants received 1 single dose of PF-04958242 0.35 mg, PF-04958242 0.6 mg, and placebo orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
  Interventions: Drug: PF-04958242; Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in treatment arm
Drug: Placebo — Administered as specified in treatment arm

SUMMARY:
This study aims to assess the safety, tolerability, and pharmacokinetics of PF-04958242 at a number of single ascending doses in healthy volunteers

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >55 kg

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2014-11-13 (Actual); Study Completion 2014-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants were assigned study treatment. All participants received the assigned PF-04958242 doses during 3 periods (6 participants each received 0.35 mg, 0.6 mg and 0.8 mg doses, respectively). Nine participants received placebo. Three participants did not complete the study and they were replaced during the conduct of the study.
Groups:
- Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg: Participants received 1 single dose of placebo, PF-04958242 0.6 mg, and PF-04958242 0.8 mg orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
- PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg: Participants received 1 single dose of PF-04958242 0.35 mg, placebo, and PF-04958242 0.8 mg orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
- PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo: Participants received 1 single dose of PF-04958242 0.35 mg, PF-04958242 0.6 mg, and placebo orally during 3 periods, respectively. There was at least a 10-day washout period between each dosing.
Period: First Intervention Period
Arm/Group | Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg | PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg | PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo
Started | 3 | 3 | 3
Completed | 2 | 2 | 2
Not Completed | 1 | 1 | 1
Not completed — No longer willing to participate | 1 | 0 | 0
Not completed — Unable to comply with study dates | 0 | 1 | 1
Period: Washout Period (at Least 10 Days)
Arm/Group | Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg | PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg | PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo
Started | 3 (One participant discontinued in the First Intervention Period and was replaced.) | 3 (One participant discontinued in the First Intervention Period and was replaced.) | 3 (One participant discontinued in the First Intervention Period and was replaced.)
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg | PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg | PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period (at Least 10 Days)
Arm/Group | Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg | PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg | PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Placebo, PF-04958242 0.6 Milligrams (mg), PF-04958242 0.8 mg | PF-04958242 0.35 mg, Placebo, PF-04958242 0.8 mg | PF-04958242 0.35 mg, PF-04958242 0.6 mg, Placebo
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Included all participants who received at least 1 dose of study treatment in any of the intervention periods
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS) Post-Baseline
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced the following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to Day 10
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Groups:
- PF-04958242 0.35 mg: All participants who received a single-dose of PF-04958242 0.35 mg capsule orally in any of the intervention periods.
- PF-04958242 0.6 mg: All participants who received a single-dose of PF-04958242 0.6 mg capsule orally in any of the intervention periods.
- PF-04958242 0.8 mg: All participants who received a single-dose of PF-04958242 0.8 mg capsule orally in any of the intervention periods.
- Placebo: All participants who received a single-dose of placebo matching capsule orally in any of the intervention periods.
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants
  Complete suicide | 0 | 0 | 0 | 0
  Suicide attempt | 0 | 0 | 0 | 0
  Preparatory acts to imminent suicidal behavior | 0 | 0 | 0 | 0
  Suicidal ideation | 0 | 0 | 0 | 0
  Self-injurious behavior, no suicidal intent | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study drug administration.
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants
  AEs | 4 | 4 | 2 | 4
  SAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], mean corpuscular hemoglobin concentration [MCHC], platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin and microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (follicle stimulating hormone [FSH], and urine drug screening).
Time Frame: Baseline up to Day 10
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants | 1 | 2 | 1 | 3

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate <40 or >120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) >=30 millimeters of mercury (mm Hg) change from baseline in same posture or SBP <90 mm Hg, diastolic blood pressure (DBP) >=20 mm Hg change from baseline in same posture or DBP <50 mm Hg. IFB = increase from baseline; DFB = decrease from baseline.
Time Frame: Baseline up to Day 10
Population: The safety analysis population included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants
  Supine SBP <90 mm Hg | 0 | 0 | 0 | 0
  Standing SBP <90 mm Hg | 0 | 0 | 0 | 0
  Supine DBP <50 mm Hg | 0 | 0 | 0 | 0
  Standing DBP <50 mm Hg | 0 | 0 | 0 | 0
  Supine Pulse Rate <40 bpm | 0 | 1 | 0 | 0
  Supine Pulse >120 bpm | 0 | 0 | 0 | 0
  Standing Pulse Rate <40 bpm | 0 | 0 | 0 | 0
  Standing Pulse Rate >140 bpm | 0 | 0 | 0 | 0
  Supine SBP >=30 mm Hg IFB | 0 | 0 | 0 | 0
  Standing SBP >=30 mm Hg IFB | 0 | 0 | 1 | 0
  Supine DBP >=20 mm Hg IFB | 0 | 0 | 0 | 0
  Standing DBP >=20 mm Hg IFB | 1 | 0 | 0 | 1
  Supine SBP >=30 mm Hg DFB | 0 | 0 | 0 | 0
  Standing SBP >=30 mm Hg DFB | 0 | 1 | 0 | 0
  Supine DBP >=20 mm Hg DFB | 0 | 0 | 0 | 0
  Standing DBP >=20 mm Hg DFB | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included pulse rate (PR) interval, QRS interval, corrected QT interval using Bazett's formula (QTcB)and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval greater than or equal to (>=)300 milliseconds (msec) or >=25% increase when baseline is greater than (>)200 msec and >=50% increase when baseline is less than or equal to (=<)200 msec; QRS interval >=140 msec or >=50% increase from baseline (IFB); and QTcF >=450 msec or >=30 msec increase. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: Baseline up to Day 10
Population: The safety analysis population included all participants who received the study medication; n=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants
  PR Interval >=300 msec | 0 | 0 | 0 | 0
  QRS Complex >=140 msec | 0 | 0 | 0 | 0
  QTcF Interval 450-<480 msec | 0 | 0 | 0 | 0
  QTcF Interval 480-<500 msec | 0 | 0 | 0 | 0
  QTcF Interval >=500 msec | 0 | 0 | 0 | 0
  QTcB Interval >=500 msec | 0 | 0 | 0 | 0
  PR Interval >=25/50% IFB | 0 | 0 | 0 | 0
  QRS Interval >=50% IFB | 0 | 0 | 0 | 0
  QTcF Interval 30-<60 msec IFB | 0 | 0 | 0 | 0
  QTcF Interval >=60 msec IFB | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The brief physical examination focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Baseline up to Day 10
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings
Description: The extended neurological examination, performed by a board certified neurologist, included observation for cerebellar (intention) tremor and for non-cerebellar tremors (eg, resting or positional), finger nose, heel shin, Romberg, tandem walking, positional and gaze evoked nystagmus, reflexes, muscle strength, cranial nerves, sensory function of upper and lower extremities. The brief neurological examination included an assessment of motor and sensory function, cranial nerves, reflexes, non-cerebellar tremor (eg, resting or positional) and cerebellar function. The assessment of cerebellar function were complemented by the Scale for Assessment and Rating of Ataxia (SARA)
Time Frame: Baseline up to Day 10
Measure: Number; unit: participants
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 9
participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: The pharmacokinetic (PK) parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 3.119 (22) | 5.602 (29) | 6.193 (24)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: The PK analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 1.29 [0.800 to 3.03] | 1.80 [0.750 to 2.00] | 1.50 [1.00 to 2.00]

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
nanograms*hours per milliliter (ng*h/mL) | 42.79 (36) | 76.00 (22) | 88.27 (23)

11. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL | 45.34 (40) | 79.34 (28) | 90.78 (26)

12. Secondary Outcome: Apparent Clearance (CL/F)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per minute (mL/min)
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
milliliters per minute (mL/min) | 128.6 (40) | 126.0 (28) | 146.9 (26)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
liters | 367.9 (45) | 327.0 (40) | 337.2 (43)

14. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 37.33 (27.170) | 34.10 (20.533) | 29.07 (14.691)

15. Secondary Outcome: Dose Normalized Cmax (Cmax[dn])
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mL/mg
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
mg/mL/mg | 8.923 (23) | 9.331 (29) | 7.745 (24)

16. Secondary Outcome: Dose Normalized AUClast (AUClast[dn])
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL/mg | 122.4 (37) | 126.6 (22) | 110.5 (24)

17. Secondary Outcome: Dose Normalized AUCinf (AUCinf[dn])
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 36, 48, 72, 96, 120, 168 and 216 hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL/mg | 129.7 (40) | 132.3 (28) | 113.6 (26)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration.
Arm/Group | PF-04958242 0.35 mg | PF-04958242 0.6 mg | PF-04958242 0.8 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-04958242 0.35 mg (N=6) | PF-04958242 0.6 mg (N=6) | PF-04958242 0.8 mg (N=6) | Placebo (N=9)
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The participants received PF-04958242 0.35 milligrams (mg), 0.6 mg and 0.8 mg instead of the proposed doses of 0.35 mg, 0.55 mg and 0.75 mg based on the review conducted after each dosing period prior to proceeding to next dosing level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.